CLINICAL TRIAL: NCT02165020
Title: Hypofractionated Radiotherapy for Prostate Cancer (62 Gy in 20 Fractions of 3.1 Gy) With Hyaluronic Acid Injection
Brief Title: Hyaluronic Acid for Hypofractionated Prostate Radiotherapy
Acronym: RPAH1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-606
Record Dates: First submitted 2014-05-05; First posted 2014-06-17 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: Prostate; Hypofractionated radiotherapy; Hyaluronic acid; Spacer; Rectum toxicity; Rectal toxicities after hypofractionated irradiation and injection of hyaluronic acid in patients with low- to intermediate-risk Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rectal toxicities after prostate hypofractionated radiotherapy (Experimental): Rectal toxicities after prostate hypofractionated radiotherapy with hyaluronic acid
  Interventions: Device: Hyaluronic acid (Macrolane VRF 30®, Q-MED)

INTERVENTIONS:
Device: Hyaluronic acid (Macrolane VRF 30®, Q-MED) — One injection of 3 to 10 cc of hyaluronic acid (Macrolane VRF 30®, Q-MED) introduced in the perirectal fat between the rectum and the prostate in connection with an ultrasound.
  The injection is performed under local anesthesia (with "Lidocaine") and ultrasound guidance, using a 16 gauge needle.

SUMMARY:
The present Phase II study aims to assess the rates of late rectal toxicities of grade ≥ 2 after hypofractionated radiotherapy of prostate cancer of 62 Gy in 20 fractions of 3.1 Gy with an injection of hyaluronic acid (HA) in the space between the rectum and the prostate. Thirty-six patients with a low- to intermediate-risk prostate cancer according to the D'Amico classification are included in the present protocol. The main characteristics of the study are that the patients benefit of a reduction of the treatment duration from 40 to 20 fractions, due to the hypofractionated irradiation, and of an injection of 3 to 10 cc of hyaluronic acid in the perirectal fat between the rectum and the prostate.

ELIGIBILITY:
Inclusion Criteria:

* age superior or equal to 18 years and inferior to 80 years.
* patient with a low- to intermediate-risk prostate cancer, according to D'Amico classification, for an exclusive irradiation.
* prostate cancer histologically proven.
* life expectancy superior to 10 years.
* Karnofsky performance status ≥ 60% (performance status ECOG 0-2).
* the patient has to be the beneficiary of a social security system or other insurance (order n° 2006-477 from April 26th 2006).
* the signed consent form.

Exclusion Criteria:

* age inferior to 18 years and ≥ 80 years;
* history of rectal surgery;
* patient who can't cooperate during the treatment;
* history of pelvic irradiation;
* history of inflammatory bowel disorder such as ulcerative colitis or the Crohn's disease;
* other current neoplasia or history of neoplasia dating from less than 5 months, excepting basal-cell carcinomas;
* patients treated with anti-neoplastic or anti-angiogenic or with other treatments used in rheumatology and which may include methotrexate (in order not to have a radiosensitizing effect);
* patients receiving anticoagulant treatment or PLAVIX;
* other undergoing study that may interfere with the present study;
* patient under legal protection measure.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-11; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with late rectal toxicities (> 3 months) of grade ≥ 2 after hypofractionated radiotherapy of prostate cancer of 62 Gy in 20 fractions of 3.1 Gy with an injection of hyaluronic acid (HA) in the space between the rectum and the prostate. | Follow-up at 3 months and 6 months after the radiotherapy and then every 6 months up to 3 years.
  Late rectal toxicities of grade ≥ 2 assessed using the CTCAE v 4.0 classification from 3 months to 3 years.

SECONDARY OUTCOMES:
Number of patients with acute rectal toxicities of all grades and of grade ≥ 2. | 3 years
  Number of patients with acute rectal toxicities of all grades and of grade ≥ 2 (using the CTCAE v 4.0), as a measure of safety and tolerability.
Tolerance of the HA injection | 3 years
  The evaluation of the tolerance of the HA injection, as a measure of safety and tolerability (using the CTCAE v 4.0).
Number of patients with acute and late toxicities, other than the rectal toxicities. | 3 years
  Number of patients with acute and late toxicities (using the CTCAE v 4.0), other than the rectal toxicities, as a measure of safety and tolerability.
The evaluation of the biochemical control | 3 years: evaluation at 3 months, 6 months and then every 6 months during the 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France